CLINICAL TRIAL: NCT01680978
Title: A SINGLE CENTER, DOUBLE-BLIND, PLACEBO-CONTROLLED, RANDOMIZED, CROSSOVER, PHASE II STUDY TO ASSESS THE EFFECT OF ALEGLITAZAR ON CARDIAC ENERGETICS AND FUNCTION IN PATIENTS WITH UNCOMPLICATED TYPE 2 DIABETES MELLITUS AND NO HISTORY OF CORONARY ARTERY DISEASE WHO ARE DRUG-NAÏVE OR TREATED WITH STABLE METFORMIN MONOTHERAPY
Brief Title: A Study to Evaluate the Effect of Aleglitazar on Cardiac Energetics and Function in Patients With Type 2 Diabetes Mellitus and no History of Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: Double
Other Study IDs: BC25445
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aleglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aleglitazar (Experimental)
  Interventions: Drug: aleglitazar
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aleglitazar — 150 mcg orally daily, 6 weeks
  Arms: Aleglitazar
Drug: placebo — orally daily, 6 weeks
  Arms: Placebo

SUMMARY:
A single center, double-blind, placebo-controlled, randomized, crossover, phase II study to assess the effect of aleglitazar on cardiac energetics and function in patients with uncomplicated type 2 diabetes mellitus and no history of coronary artery disease who are drug-naïve or treated with stable metformin. Eligible patients will receive either 150 mcg aleglitazar or placebo orally daily for 6 weeks. After a washout period of 6 weeks, patients will cross over to the treatment not yet received.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 40 to 70 years of age (inclusive) at screening
* Patients with Type 2 diabetes mellitus diagnosed at least 12 weeks before screening and either drug-naïve or treated with stable metformin monotherapy for at least 12 weeks prior to screening
* HbA1c >/= 7 % and </= 9% at screening
* Absence of history of coronary artery disease

Exclusion Criteria:

* Diagnosis or history of Type 1 diabetes mellitus, diabetes resulting from pancreatic injury, or secondary forms of diabetes
* Current treatment with fibrates, thiazolidinediones, or insulin
* Prior intolerance to thiazolidinediones and/or fibrates
* Clinically significant liver disease or impaired liver function
* Know chronic diabetic complications (i.e. retinopathy, neuropathy, nephropathy)
* Symptomatic congestive heart failure classified as NYHA class II-IV
* Diagnosed and/or treated malignancy within the past 5 years, except for treated basal cell skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer
* Contraindications to MRI, or inability to tolerate MRI scanning

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cardiac energetics: Change in PCr/ATP ratio using phosphorus magnetic resonance spectroscopy (MRS) | from baseline to Week 6

SECONDARY OUTCOMES:
Change in left ventricular diastolic function measured by mitral inflow, tissue Doppler Imaging and magnetic resonance imaging (MRI) | from baseline to Week 6
Change in cardiac/hepatic triglyceride content assessed my MRS | from baseline to Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Oxford, United Kingdom